CLINICAL TRIAL: NCT04068246
Title: The AMPK Modulator Metformin as a Novel Adjunct to Conventional Therapy in Rheumatoid Arthritis Patients: A Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled Trial.
Brief Title: The AMPK Modulator Metformin as a Novel Adjunct to Conventional Therapy in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, PhD., Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMRR-8-2019
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (Placebo Comparator): patients will receive the standard therapy (methotrexate) plus placebo tablets
  Interventions: Drug: Placebo
- Metformin group (Experimental): patients will receive the standard therapy plus 1 g metformin daily.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 1000 mg of Metformin table taken orally daily plus Methotrexate 7.5 mg weekly
  Arms: Metformin group
Drug: Placebo — Placebo tablet plus plus Methotrexate 7.5 mg weekly
  Arms: Control group

SUMMARY:
Metformin, a traditional antidiabetic medication, exerts glucose lowering effects by activating AMP-activated protein kinase (AMPK), a critical enzyme involved in the lipid and glucose metabolism. In addition to the antidiabetic effect, metformin has been shown to inhibit Lipopolysaccharide-Induced Inflammation (LPS)-induced inflammation by suppress NF-κB production, which is also regulated by AMPK. These regulatory effects of AMPK on the inflammation, immune and fibroblast-like synovial cells have prompted the investigation on the effects of metformin on rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, multisystem inflammatory disorder of unknown etiology. It is characterized by polyarthritis and systemic inflammation. The inflammation in the hyperplastic synovium can destruct the structure of affected joints. Although the exact molecular mechanism underlying the pathogenesis of RA remains unknown, it is suggested that T helper cell (Th) 17 plays a central role. Interleukin (IL)-17, mostly secreted by Th17, has synergistic effects with tumor necrosis factor- (TNF-α), IL-1β and IL-6 in cases of RA. Metformin, a traditional antidiabetic medication, exerts glucose lowering effects by activating AMP-activated protein kinase (AMPK), a critical enzyme involved in the lipid and glucose metabolism. In addition to the antidiabetic effect, metformin has been shown to inhibit Lipopolysaccharide-Induced Inflammation (LPS)-induced inflammation by suppress NF-κB production, which is also regulated by AMPK . In addition, metformin activated AMPK may inhibit mammalian target of rapamycin (mTOR), which then regulate the differentiation of T cells in vitro and in vivo. In particular, AMPK has been reported to be associated with the inhibition of TH17 cells through suppressing the phosphorylation of mTOR and its downstream signal transducers, suggesting the therapeutic potential of AMPK agonists. Besides the imbalance between Th17 cells and Treg cells is responsible for the chronic inflammation in RA, synovium hyperplasia also plays a central role in the joint destruction. It has been reported that rapamycin, an inhibitor of mTOR, is able to significantly reduce fibroblastlike synovial cell invasion in RA via suppressing mTOR signaling pathway. These regulatory effects of AMPK on the inflammation, immune and fibroblast-like synovial cells have prompted the investigation on the effects of metformin on rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active rheumatoid arthritis based on DAS28 score. Patients received the standard therapy (i.e. one or more conventional DMARDs) for at least three months.

Exclusion Criteria:

* Known hypersensitivity to metformin.
* Patients who have a prior diagnosis with diabetes mellitus.
* Patients receive metformin for any other indications.
* Patients with congestive heart failure.
* Patients with a history of myocardial infarction.
* Patients with severe anemia.
* Patients with active infections or other inflammatory diseases.
* Patients receiving biological therapy.
* Pregnancy or lactation.
* Patients with impaired liver functions.
* Patients with impaired kidney functions (serum creatinine concentrations ≥1.5 and ≥1.4 mg/dL in males and females respectively).
* Patients with malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
ACR 20% improvement criteria (ACR20) response rate | week 12
  based on tender and swollen joint counts, patient's assessment of pain, patient and physician global assessment of arthritis, Health Assessment Questionnaire Disability Index (HAQ DI), and CRP level
ACR50 & ACR70 response rate | week 12
  based on tender and swollen joint counts, patient's assessment of pain, patient and physician global assessment of arthritis, Health Assessment Questionnaire Disability Index (HAQ DI), and CRP level
Disease activity scale in 28 joints (DAS-28) | week 12
  Scale assessing severity of rheumatoid arthritis based on number of tender, swollen joints, erythrocyte sedimentation rate (ESR) levels, and patient self-assessment of his condition (global health assessment). Whereas "28" describes the number of different joints including in the measurement: proximal interphalangeal joints (10 joints), metacarpophalangeal joints (10), wrists (2), elbows (2), shoulders (2), knees (2).

SECONDARY OUTCOMES:
the Short Form 36 (SF-36) Health Survey | week 12
  both the physical component score [PCS] and the mental component score [MCS])
HAQ-DI (Health Assessment Score- Disability index) | week 12
  HAQ-DI (Health Assessment Score- Disability index), in which patients are asked to rate their capacity to perform 20 activities of daily living (ADL). Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section
AMPK expression | at baseline and at week 12
  AMPK expression in synovium or serum
IGF-IR expression | at baseline and at week 12
  IGF-IR expression in Blood
TNF-α | at baseline and at week 12
  Serum level Tumor necrosis factor- alpha (TNF-α)
TGF-Beta1 | at baseline and at week 12
  Serum level tissue growth factor beta 1
Inteleukins | at baseline and at week 12
  Serum levels of Interleukins (IL) IL-17, IL-1β , IL-6 & IL-10
CRP | at baseline and at week 12
  Serum level of C-reactive protein (CRP)
Drug Adverse effects | 3 months
  Adverse effect incidence: adverse effect will be reported by patients or their caregivers and recorded by investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Abdallah MS, Alarfaj SJ, Saif DS, El-Naggar ME, Elsokary MA, Elsawah HK, Abdelsattar Zaki S, Wahsh EA, Abo Mansour HE, Mosalam EM. The AMPK modulator metformin as adjunct to methotrexate in patients with rheumatoid arthritis: A proof-of-concept, randomized, double-blind, placebo-controlled trial. Int Immunopharmacol. 2021 Jun;95:107575. doi: 10.1016/j.intimp.2021.107575. Epub 2021 Mar 24. PMID 33773207
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33773207/